CLINICAL TRIAL: NCT01579448
Title: A Open Labeled Controlled Trial to Evaluate the Immune Response of a Boosting Regimen With Shanchol™, a Killed Whole Cell Oral Cholera Vaccine (WC-OCV), in Previously Immunized Adults and Children in Eastern Kolkata, India
Brief Title: Evaluation of a Boosting Regimen With Oral Cholera Vaccine
Acronym: Boost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sachin Desai (Other)
Collaborators: National Institute of Cholera and Enteric Diseases, India (Other); Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor-Investigator, Sachin Desai, ASSOCIATE RESEARCH SCIENTIST, International Vaccine Institute
Organization: International Vaccine Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR-WC-11
Record Dates: First submitted 2012-04-11; First posted 2012-04-18 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Cholera
Keywords: killed oral cholera vaccine; boosting vaccine regimen; safety and immunogenicity
MeSH Terms: conditions — Cholera | interventions — shanchol; Cholera Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine to past vaccinated participants (Experimental): The first arm includes subjects, who were immunized with two Shanchol™ doses, five years prior. In this study, arm one will receive one Shanchol™ booster dose at baseline and one booster dose on day fourteen.
  Interventions: Biological: Shanchol™, oral cholera vaccine
- Vaccine to past placebo recipients (Active Comparator): The second arm includes subjects, who received two placebo doses, five years prior. Arm two will receive a primary immunization series consisting of one Shanchol™ dose at baseline and one at day fourteen
  Interventions: Biological: Shanchol™, killed, whole cell, bivalent, oral cholera vaccine
- No intervention to past placebo recipients (Placebo Comparator): The third arm includes subjects, who received two placebo doses, five years prior. This third arm will not receive any intervention and will serve to represent a baseline immune response by vaccine naïve individuals exposed to natural exposure.
  Interventions: Other: no intervention

INTERVENTIONS:
Biological: Shanchol™, oral cholera vaccine — This killed, whole cell, bivalent vaccine will be presented as a creamish white suspension. Upon storage, a white sediment and clear supernatant may be observed. The recommended dose (1.5ml) of the vaccine must be administered orally. The primary vaccination schedule consists of two doses given at an interval of two weeks. After vigorous shaking of the vial, 1.5 ml should be poured into the mouth of the recipient, followed by water ad libitum. The vaccine can alternatively be administered with a disposable syringe (without needle) after removing the contents from the vial and squirted into the mouth of the recipient.
  Vaccine is administered in 1.5 mL vials by mouth in 2 doses, given 2 weeks apart. The vaccine appears as a creamy white suspension.
  Arms: Vaccine to past vaccinated participants
Biological: Shanchol™, killed, whole cell, bivalent, oral cholera vaccine — This killed, whole cell, bivalent vaccine will be presented as a creamish white suspension. Upon storage, a white sediment and clear supernatant may be observed. The recommended dose (1.5ml) of the vaccine must be administered orally. The primary vaccination schedule consists of two doses given at an interval of two weeks. After vigorous shaking of the vial, 1.5 ml should be poured into the mouth of the recipient, followed by water ad libitum. The vaccine can alternatively be administered with a disposable syringe (without needle) after removing the contents from the vial and squirted into the mouth of the recipient.
  Vaccine is administered in 1.5 mL vials by mouth in 2 doses, given 2 weeks apart. The vaccine appears as a creamy white suspension.
  Arms: Vaccine to past placebo recipients
Other: no intervention — No intervention will be given to this arm of past placebo recipients. To ensure that boosting was not due to natural exposure to Vibrio cholera, we will compare subjects in the boosting arm to this no intervention arm.
  Arms: No intervention to past placebo recipients

SUMMARY:
Data demonstrates that Shanchol™ (killed bivalent oral cholera vaccine) provides protection over 3 years and data regarding the protective efficacy over five years is anticipated for 2012. Regardless at the end of five years, it may still be necessary to provide a booster dose or reimmunize with two doses to maintain protection in previously immunized populations. This study examines the immune protection and safety of providing a one and two dose boosting regimen of Shanchol™ given five years after the initial dose.

ELIGIBILITY:
Inclusion Criteria:

All subjects must be presently enrolled in the Phase 3 NICED RCT of Shanchol™ and satisfy the following criteria at study entry:

1. Male or female adults aged 6 years and above, who are available for follow-up visits and specimen collection.

   * The subject should be able to continue in the study for the next 6 weeks
   * The subject (or parent/guardian) should be willing to provide 3 blood samples
2. Written informed consent obtained from the subjects or their parents/guardians, and written assent obtained from children aged 12 - 17 years.
3. Healthy subjects as determined by:

   * Medical history
   * Physical examination
   * Clinical judgment of the investigator

Exclusion Criteria:

1. individuals who are too weak to get out of bed to receive the vaccine
2. pregnant women (identified through verbal screening)
3. those less than 6 years of age
4. Receipt of cholera vaccine following 2009 (time of licensure and availability of Shanchol™ in India)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity provided by a two dose boosting regimen of Shanchol™ | 28 days
  To determine whether two doses of Shanchol™ administered to a previously immunized cohort elicits similar immune responses (greater than fourfold rise in serum vibriocidal antibody titers through IgM) to those achieved by a primary immunization series in an unimmunized cohort stratified by age (6-14 and ≥15 years old),

SECONDARY OUTCOMES:
Immunogenicity provided by a one dose boosting regimen of Shanchol™ | 28 days
  To determine if a one dose booster regimen of Shanchol™ administered to a previously immunized cohort can elicit similar immune responses (through serum IgM) to those achieved by primary immunization in an unimmunized cohort stratified by age (6-14 and ≥15 years old)
Rises in serum IgA and IgG following boosting regimens | 28 days
  Measure rises in serum IgA and IgG as an adjunct measure of immunogenic response to the Shanchol™ boosting regimens
Proportion of subjects with adverse events | 42 days
  To confirm the safety of one and two dose boosting regimens Shanchol™ in healthy, non-pregnant subjects stratified by age within 28 days following dosing in each intervention group. Screening for number of adverse events (AEs)and severe adverse events (SAEs) will done on all study visits. Adverse events screened for include: diarrhea, fever, vomiting, abdominal pain, itching, rash, nausea, weakness, cough, vertigo, and dryness of mouth. SAEs are those which are incapacitating, preventing normal activities, including death and hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Kanungo, MBBS, Principal Investigator — National Institute of Cholera and Enteric Diseases, India
Locations (1):
- National Institute of Cholera and Enteric Diseases, Kolkata, West Bengal, India